CLINICAL TRIAL: NCT00544323
Title: Alveolar Bone Loss Around 3 Different Designs of Dental Implant: Prospective Comparative Clinical Trail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: cobiHMO
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2007-10

CONDITIONS: Alveolar Bone Loss
Keywords: alveolar bone; radiographic alveolar bone changes around oral implants of various designs 12 m post loading
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: oral implant

SUMMARY:
comparison of alveolar bone resorbtion/ changes for a period of 12 month post loading of different designs and brands of oral implants. in this study, a comparison between straumann SLA-active implants to MIS Mistral and Mistral -X implants.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* >18Y
* consent
* posterior mandibular missing teeth

Exclusion Criteria:

* chronic illness: diabetes, artheritis
* women: pregnancy, lactation
* non consent
* alcohol consumption
* smoking >10 p day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2007-11

PRIMARY OUTCOMES:
radiographic changes in the alveolar bone height around the oral implant till 12 m post loading | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lior Shapira Prof, Study Chair — Hadassah Medical Organization
Locations (1):
- Hadassah medical center, school of dentistry, Jerusalem, Israel